CLINICAL TRIAL: NCT03631628
Title: A Randomized Controlled Clinical Trial of Upper Limb Training with Mirror Therapy (MT) and Bilateral Transcutaneous Electrical Nerve Stimulation (Bi-TENS) to Improve Upper Limb Motor Functions in Patients with Stroke
Brief Title: Upper Limb Mirror Therapy with Bilateral Transcutaneous Electrical Nerve Stimulation to Improve Upper Limb Functions in Patients with Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Shamay Ng, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019_MT_TENS_UL
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MT+ Bilateral TENS (Experimental): All subjects will undergo 16 sessions of treatment (2 times per week, for 8 weeks). Subjects will receive 1.5 hours rehabilitation program: 30 minutes of MT+bilateral TENS and 1 hour conventional training of standardized upper limb training.
  Interventions: Device: Bilateral Transcutaneous electrical nerve stimulation (Bi-TENS); Behavioral: Mirror Therapy (MT); Behavioral: Conventional Rehabilitation Program
- sham-MT+ Bilateral TENS (Placebo Comparator): All subjects will undergo 16 sessions of treatment (2 times per week, for 8 weeks). Subjects will receive 1.5 hours rehabilitation program: 30 minutes of sham-MT+bilateral TENS and 1 hour conventional training of standardized upper limb training.
  Interventions: Device: Bilateral Transcutaneous electrical nerve stimulation (Bi-TENS); Behavioral: sham-Mirror Therapy (sham-MT); Behavioral: Conventional Rehabilitation Program

INTERVENTIONS:
Device: Bilateral Transcutaneous electrical nerve stimulation (Bi-TENS) — The stimulator is a 120z Dual-Channel TENS Unit (ITO Physiotherapy & Rehabilittaion, Co, Ltd, Tokyo, Japan). The TENS stimulation will be at 100 Hz, with 0.2 ms square pulses at an intensity of twice the sensory threshold (defined as the minimum intensity at which subject reported feeling a tingling sensation and below the motor threshold as indicated by the absence of muscle twitching, to provide sensory stimulation to both paretic and intact arms. Two pairs of disposable surface electrodes will be applied over the median nerve from the carpal tunnel to the flexor digitorum superficialis and the superficial radial nerve from the extensor pollicis longus to the extensor digitorum communis, with the cathode on the proximal site, and the anode on the distal site.
Behavioral: Mirror Therapy (MT) — A customised angle-adjustable frame with a mirror board will be used. All subjects are instructed to perform
  1. Elbow flexion and extension exercise
  2. Forearm pronation and supination exercise
  3. Wrist flexion and extension exercise
  4. Wrist radial and ulnar deviation exercise
  5. Fingers opposition exercise
  6. Gripping exercise
  The subject will complete bilaterally upper limb exercises during the 30 minutes period.
  Intact arm will be placed in front of mirror, and paretic arm will be placed behind the mirror.
  Joints involved will be flexed and extended in full available range in sitting positon, in order to improve the active control of elbow joint, wrist joint and all fingers joint respectively.
  Participants will be encouraged to focus on the image of intact arm when performing upper limb exercises bilaterally.
  Arms: MT+ Bilateral TENS
Behavioral: sham-Mirror Therapy (sham-MT) — A customised angle-adjustable frame with a mirror board will be used while the reflecting surface of the mirror was covered with paper. All subjects are instructed to perform
  1. Elbow flexion and extension exercise
  2. Forearm pronation and supination exercise
  3. Wrist flexion and extension exercise
  4. Wrist radial and ulnar deviation exercise
  5. Fingers opposition exercise
  6. Gripping exercise
  The subject will complete bilaterally upper limb exercises during the 30 minutes period.
  Intact arm will be placed in front of covered mirror, and paretic arm will be placed behind the covered mirror.
  Joints involved will be flexed and extended in full available range in sitting positon, in order to improve the active control of elbow joint, wrist joint and all fingers joint respectively.
  Arms: sham-MT+ Bilateral TENS
Behavioral: Conventional Rehabilitation Program — Standardized upper limb training

SUMMARY:
This study compare the effectiveness of 2 rehabilitation programmes that use (1) MT with Bilateral TENS (Bi-TENS), (2) sham-MT with Bi-TENS (Bi-TENS), respectively, in addition to conventional rehabilitation of standardized upper limb training, in improving upper limb motor functions, activities of daily living, community integration, and quality of life in patients with stroke.

DETAILED DESCRIPTION:
The principal aim of the proposed study will be to demonstrate whether MT with Bi-TENS is more effective than sham-MT with Bi-TENS in improving upper limb motor functions, activities of daily living, community integration and quality of life in patients with stroke.

The null hypothesis will be that MT with Bi-TENS is not significantly different from sham-MT with Bi-TENS in improving upper limb motor functions, activities of daily living, community integration, and quality of life in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

1. have been diagnosed with ischemic brain injury or intracerebral hemorrhage by MRI or computed tomography within three weeks to 10 years after the first onset of stroke;
2. have volitional control of the non-paretic arm, and at least minimal antigravity movement in the shoulder of the paretic arm;
3. have at least 5 degrees in wrist extension of the paretic arm in the antigravity position
4. are able to score > 6 of 10 of abbreviated Mental Test;
5. are able to follow instruction and give informed consent of the study.

Exclusion Criteria:

1. Have any additional medical, cardiovascular and orthopedic condition that would hinder the proper assessment and treatment;
2. Use cardiac pacemakers;
3. Have receptive dysphasia;
4. Have a significant upper limb peripheral neuropathy (e.g., diabetic polyneuropathy);
5. Have severe shoulder, elbow, wrist or finger contractures that would preclude a passive range of motions of the arm;
6. Have skin allergy that would prevent electrical stimulation;
7. Are involved in drug studies or other clinical trials.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment of Upper Extremity (FMA-UE) - baseline | Baseline (0 week)
  The FMA-UE will be used to evaluate the severity of motor impairment in the paretic upper extremity. The performance of 33 tasks will be assessed using a three-point ordinal scale (0 to 2), with a maximum score of 66. The FMA-UE will assess voluntary movement, reflex activity, grasp, and coordination of the upper extremity, and has a high inter-rater reliability (r=0.99) in patients with stroke. A higher scale score indicates a less severe motor impairment.
Fugl-Meyer Assessment of Upper Extremity (FMA-UE) - midterm | 4 weeks
  The FMA-UE will be used to evaluate the severity of motor impairment in the paretic upper extremity. The performance of 33 tasks will be assessed using a three-point ordinal scale (0 to 2), with a maximum score of 66. The FMA-UE will assess voluntary movement, reflex activity, grasp, and coordination of the upper extremity, and has a high inter-rater reliability (r=0.99) in patients with stroke. A higher scale score indicates a less severe motor impairment.
Fugl-Meyer Assessment of Upper Extremity (FMA-UE) - post-training | 8 weeks
  The FMA-UE will be used to evaluate the severity of motor impairment in the paretic upper extremity. The performance of 33 tasks will be assessed using a three-point ordinal scale (0 to 2), with a maximum score of 66. The FMA-UE will assess voluntary movement, reflex activity, grasp, and coordination of the upper extremity, and has a high inter-rater reliability (r=0.99) in patients with stroke. A higher scale score indicates a less severe motor impairment.
Fugl-Meyer Assessment of Upper Extremity (FMA-UE) - followup | 12 weeks
  The FMA-UE will be used to evaluate the severity of motor impairment in the paretic upper extremity. The performance of 33 tasks will be assessed using a three-point ordinal scale (0 to 2), with a maximum score of 66. The FMA-UE will assess voluntary movement, reflex activity, grasp, and coordination of the upper extremity, and has a high inter-rater reliability (r=0.99) in patients with stroke. A higher scale score indicates a less severe motor impairment.
Wolf Motor Function Test (WMFT) - baseline | Baseline (0 week)
  Upper limb function will be assessed by the WMFT, which comprises two items of strength-based tasks, and 15 items of function-based tasks. The two strength-based tasks will be measured by weight lift and grip strength. The 15 function-based tasks will be assessed by the time taken to complete each task (in seconds), and the quality rating of the use of the paretic hand in attempting each task (graded 0 to 5). The scores for the 15 tasks will be summed and then averaged to yield the mean functional ability score. The WMFT has a high inter-rater reliability (ICC=0.97) and test-retest reliability for time scores (ICC=0.95). A higher score indicates a better hand function.
Wolf Motor Function Test (WMFT) - midterm | 4 weeks
  Upper limb function will be assessed by the WMFT, which comprises two items of strength-based tasks, and 15 items of function-based tasks. The two strength-based tasks will be measured by weight lift and grip strength. The 15 function-based tasks will be assessed by the time taken to complete each task (in seconds), and the quality rating of the use of the paretic hand in attempting each task (graded 0 to 5). The scores for the 15 tasks will be summed and then averaged to yield the mean functional ability score. The WMFT has a high inter-rater reliability (ICC=0.97) and test-retest reliability for time scores (ICC=0.95). A higher score indicates a better hand function.
Wolf Motor Function Test (WMFT) - post-training | 8 weeks
  Upper limb function will be assessed by the WMFT, which comprises two items of strength-based tasks, and 15 items of function-based tasks. The two strength-based tasks will be measured by weight lift and grip strength. The 15 function-based tasks will be assessed by the time taken to complete each task (in seconds), and the quality rating of the use of the paretic hand in attempting each task (graded 0 to 5). The scores for the 15 tasks will be summed and then averaged to yield the mean functional ability score. The WMFT has a high inter-rater reliability (ICC=0.97) and test-retest reliability for time scores (ICC=0.95). A higher score indicates a better hand function.
Wolf Motor Function Test (WMFT) - followup | 12 weeks
  Upper limb function will be assessed by the WMFT, which comprises two items of strength-based tasks, and 15 items of function-based tasks. The two strength-based tasks will be measured by weight lift and grip strength. The 15 function-based tasks will be assessed by the time taken to complete each task (in seconds), and the quality rating of the use of the paretic hand in attempting each task (graded 0 to 5). The scores for the 15 tasks will be summed and then averaged to yield the mean functional ability score. The WMFT has a high inter-rater reliability (ICC=0.97) and test-retest reliability for time scores (ICC=0.95). A higher score indicates a better hand function.

SECONDARY OUTCOMES:
Grip Strength - baseline | Baseline (0 week)
  Grip strength of both the paretic and intact hands will be measured using the Jamar dynamometer (Sammons Preston Rolyan, Bolingbrook, IL, USA) with standardized positioning and instructions recommended by the American Society of Hand Therapist. All subjects will be required to squeeze the dynamometer as hard as possible for 5 s for three trials. The force generated (in kilograms) in all three trials will be recorded and averaged for data analysis. The measurement of grip strength with the dynamometer has a high test-retest reliability (r=0.88-0.93) and inter-rater reliability (r=0.99).
Grip Strength - midterm | 4 weeks
  Grip strength of both the paretic and intact hands will be measured using the Jamar dynamometer (Sammons Preston Rolyan, Bolingbrook, IL, USA) with standardized positioning and instructions recommended by the American Society of Hand Therapist. All subjects will be required to squeeze the dynamometer as hard as possible for 5 s for three trials. The force generated (in kilograms) in all three trials will be recorded and averaged for data analysis. The measurement of grip strength with the dynamometer has a high test-retest reliability (r=0.88-0.93) and inter-rater reliability (r=0.99).
Grip Strength - post-training | 8 weeks
  Grip strength of both the paretic and intact hands will be measured using the Jamar dynamometer (Sammons Preston Rolyan, Bolingbrook, IL, USA) with standardized positioning and instructions recommended by the American Society of Hand Therapist. All subjects will be required to squeeze the dynamometer as hard as possible for 5 s for three trials. The force generated (in kilograms) in all three trials will be recorded and averaged for data analysis. The measurement of grip strength with the dynamometer has a high test-retest reliability (r=0.88-0.93) and inter-rater reliability (r=0.99).
Grip Strength - followup | 12 weeks
  Grip strength of both the paretic and intact hands will be measured using the Jamar dynamometer (Sammons Preston Rolyan, Bolingbrook, IL, USA) with standardized positioning and instructions recommended by the American Society of Hand Therapist. All subjects will be required to squeeze the dynamometer as hard as possible for 5 s for three trials. The force generated (in kilograms) in all three trials will be recorded and averaged for data analysis. The measurement of grip strength with the dynamometer has a high test-retest reliability (r=0.88-0.93) and inter-rater reliability (r=0.99).
Jacket Test - baseline | Baseline (0 week)
  The Jacket Test will be used to assess the stroke patients' upper limb proficiency in putting on and removing a long-sleeved jacket. The test will be performed in the standing position. The total time will be calculated by stopwatch as the sum of time to put on and take off clothes. The Jacket Test will be tested three times. Three trials of the Jacket Test time will be collected and averaged for data analysis. This test has excellent intra-rater, inter-rater and test-retest reliability (ICC = 0.781 - 1.000) in people with stroke.
Jacket Test - midterm | 4 weeks
  The Jacket Test will be used to assess the stroke patients' upper limb proficiency in putting on and removing a long-sleeved jacket. The test will be performed in the standing position. The total time will be calculated by stopwatch as the sum of time to put on and take off clothes. The Jacket Test will be tested three times. Three trials of the Jacket Test time will be collected and averaged for data analysis. This test has excellent intra-rater, inter-rater and test-retest reliability (ICC = 0.781 - 1.000) in people with stroke.
Jacket Test - post-training | 8 weeks
  The Jacket Test will be used to assess the stroke patients' upper limb proficiency in putting on and removing a long-sleeved jacket. The test will be performed in the standing position. The total time will be calculated by stopwatch as the sum of time to put on and take off clothes. The Jacket Test will be tested three times. Three trials of the Jacket Test time will be collected and averaged for data analysis. This test has excellent intra-rater, inter-rater and test-retest reliability (ICC = 0.781 - 1.000) in people with stroke.
Jacket Test - followup | 12 weeks
  The Jacket Test will be used to assess the stroke patients' upper limb proficiency in putting on and removing a long-sleeved jacket. The test will be performed in the standing position. The total time will be calculated by stopwatch as the sum of time to put on and take off clothes. The Jacket Test will be tested three times. Three trials of the Jacket Test time will be collected and averaged for data analysis. This test has excellent intra-rater, inter-rater and test-retest reliability (ICC = 0.781 - 1.000) in people with stroke.
Upper Extremity Functional Index (UEFI) - baseline | Baseline (0 week)
  The UEFI will be used to evaluate the upper extremity functional recovery among community-dwelling people with chronic stroke. UEFI contains 15 items with five patient-reported difficulty level (0 to 4), with a maximum score of 59. The UEFI has a good test-retest resliability (ICC = 0.87) and excellent internal consistency (Cronbach's α = 0.922) in people with chronic stroke. A higher score indicates a higher upper extremity functional recovery in people with chronic stroke.
Upper Extremity Functional Index (UEFI) - midterm | 4 weeks
  The UEFI will be used to evaluate the upper extremity functional recovery among community-dwelling people with chronic stroke. UEFI contains 15 items with five patient-reported difficulty level (0 to 4), with a maximum score of 59. The UEFI has a good test-retest resliability (ICC = 0.87) and excellent internal consistency (Cronbach's α = 0.922) in people with chronic stroke. A higher score indicates a higher upper extremity functional recovery in people with chronic stroke.
Upper Extremity Functional Index (UEFI) - post-training | 8 weeks
  The UEFI will be used to evaluate the upper extremity functional recovery among community-dwelling people with chronic stroke. UEFI contains 15 items with five patient-reported difficulty level (0 to 4), with a maximum score of 59. The UEFI has a good test-retest resliability (ICC = 0.87) and excellent internal consistency (Cronbach's α = 0.922) in people with chronic stroke. A higher score indicates a higher upper extremity functional recovery in people with chronic stroke.
Upper Extremity Functional Index (UEFI) - followup | 12 weeks
  The UEFI will be used to evaluate the upper extremity functional recovery among community-dwelling people with chronic stroke. UEFI contains 15 items with five patient-reported difficulty level (0 to 4), with a maximum score of 59. The UEFI has a good test-retest resliability (ICC = 0.87) and excellent internal consistency (Cronbach's α = 0.922) in people with chronic stroke. A higher score indicates a higher upper extremity functional recovery in people with chronic stroke.
Motor Activity Log (MAL) - baseline | Baseline (0 week)
  The MAL questionnaire will be used to assess how frequently and how well a person uses the paretic upper limb in 30 activities of daily life in a semi-structured interview. Based on a six-point ordinal scale, subjects will be required to rate (1) the amount of use (AOU), and (2) the quality of movement (QOM) when performing these 30 tasks in real life situations. The AOU and QOM scores will be summed and averaged to yield a single MAL score for each subject. The MAL has high internal consistency (Cronbach alpha > 0.88), and reasonable construct validity (Spearman r=0.63) in patients with stroke, and the Chinese version of the MAL will be used in this study. A higher score indicates a better use of the affected hand in daily life.
Motor Activity Log (MAL) - midterm | 4 weeks
  The MAL questionnaire will be used to assess how frequently and how well a person uses the paretic upper limb in 30 activities of daily life in a semi-structured interview. Based on a six-point ordinal scale, subjects will be required to rate (1) the amount of use (AOU), and (2) the quality of movement (QOM) when performing these 30 tasks in real life situations. The AOU and QOM scores will be summed and averaged to yield a single MAL score for each subject. The MAL has high internal consistency (Cronbach alpha > 0.88), and reasonable construct validity (Spearman r=0.63) in patients with stroke, and the Chinese version of the MAL will be used in this study. A higher score indicates a better use of the affected hand in daily life.
Motor Activity Log (MAL) - post-training | 8 weeks
  The MAL questionnaire will be used to assess how frequently and how well a person uses the paretic upper limb in 30 activities of daily life in a semi-structured interview. Based on a six-point ordinal scale, subjects will be required to rate (1) the amount of use (AOU), and (2) the quality of movement (QOM) when performing these 30 tasks in real life situations. The AOU and QOM scores will be summed and averaged to yield a single MAL score for each subject. The MAL has high internal consistency (Cronbach alpha > 0.88), and reasonable construct validity (Spearman r=0.63) in patients with stroke, and the Chinese version of the MAL will be used in this study. A higher score indicates a better use of the affected hand in daily life.
- Motor Activity Log (MAL) - followup | 12 weeks
  The MAL questionnaire will be used to assess how frequently and how well a person uses the paretic upper limb in 30 activities of daily life in a semi-structured interview. Based on a six-point ordinal scale, subjects will be required to rate (1) the amount of use (AOU), and (2) the quality of movement (QOM) when performing these 30 tasks in real life situations. The AOU and QOM scores will be summed and averaged to yield a single MAL score for each subject. The MAL has high internal consistency (Cronbach alpha > 0.88), and reasonable construct validity (Spearman r=0.63) in patients with stroke, and the Chinese version of the MAL will be used in this study. A higher score indicates a better use of the affected hand in daily life.
Stroke Impact Scale (SIS) - baseline | Baseline (0 week)
  SIS will be used to evaluate the health-related quality of life in stroke survivors. The SIS is a 59-item questionnaire which consists of 8 domains: Strength (4 items), memory and thinking (7 items), emotion (9 items), communication (7 items), ADL (10 items), mobility (9 items), hand function (5 items), and participation (8 items). Responses to each item will be based on a 5-point Likert scale that ask participants to score their level of difficulty with a task over the previous 2 weeks. Items from strength, ADL, mobility and hand function domains can be combined to create a composite physical functioning score. Scores for each domain are transformed into a score out of 100 using the formula: [(mean domain score-1)/(5-1)]*100. A higher score is indicative of better self-perceived health. The SIS has demonstrated validity and reliability for assessing health-related QoL.
Stroke Impact Scale (SIS) - midterm | 4 weeks
  SIS will be used to evaluate the health-related quality of life in stroke survivors. The SIS is a 59-item questionnaire which consists of 8 domains: Strength (4 items), memory and thinking (7 items), emotion (9 items), communication (7 items), ADL (10 items), mobility (9 items), hand function (5 items), and participation (8 items). Responses to each item will be based on a 5-point Likert scale that ask participants to score their level of difficulty with a task over the previous 2 weeks. Items from strength, ADL, mobility and hand function domains can be combined to create a composite physical functioning score. Scores for each domain are transformed into a score out of 100 using the formula: [(mean domain score-1)/(5-1)]*100. A higher score is indicative of better self-perceived health. The SIS has demonstrated validity and reliability for assessing health-related QoL.
Stroke Impact Scale (SIS) - post-training | 8 weeks
  SIS will be used to evaluate the health-related quality of life in stroke survivors. The SIS is a 59-item questionnaire which consists of 8 domains: Strength (4 items), memory and thinking (7 items), emotion (9 items), communication (7 items), ADL (10 items), mobility (9 items), hand function (5 items), and participation (8 items). Responses to each item will be based on a 5-point Likert scale that ask participants to score their level of difficulty with a task over the previous 2 weeks. Items from strength, ADL, mobility and hand function domains can be combined to create a composite physical functioning score. Scores for each domain are transformed into a score out of 100 using the formula: [(mean domain score-1)/(5-1)]*100. A higher score is indicative of better self-perceived health. The SIS has demonstrated validity and reliability for assessing health-related QoL.
Stroke Impact Scale (SIS) - followup | 12 weeks
  SIS will be used to evaluate the health-related quality of life in stroke survivors. The SIS is a 59-item questionnaire which consists of 8 domains: Strength (4 items), memory and thinking (7 items), emotion (9 items), communication (7 items), ADL (10 items), mobility (9 items), hand function (5 items), and participation (8 items). Responses to each item will be based on a 5-point Likert scale that ask participants to score their level of difficulty with a task over the previous 2 weeks. Items from strength, ADL, mobility and hand function domains can be combined to create a composite physical functioning score. Scores for each domain are transformed into a score out of 100 using the formula: [(mean domain score-1)/(5-1)]*100. A higher score is indicative of better self-perceived health. The SIS has demonstrated validity and reliability for assessing health-related QoL.
Community Integration Questionnaire (CIM) - baseline | Baseline (0 week)
  The level of community integration will be assessed by the Cantonese version of Community Integration Measures (CIM-C). The CIM is a client-centred questionnaire with 10 items; each item solicits a rating on a 5-point scale for a total score from 10 to 50. The CIM-C has demonstrated good internal consistency (Cronbach α, 0.84) and reliability (ICC, 0.84). A higher score indicates a higher level of community integration.
Community Integration Questionnaire (CIM) - midterm | 4 weeks
  The level of community integration will be assessed by the Cantonese version of Community Integration Measures (CIM-C). The CIM is a client-centred questionnaire with 10 items; each item solicits a rating on a 5-point scale for a total score from 10 to 50. The CIM-C has demonstrated good internal consistency (Cronbach α, 0.84) and reliability (ICC, 0.84). A higher score indicates a higher level of community integration.
Community Integration Questionnaire (CIM) - post-training | 8 weeks
  The level of community integration will be assessed by the Cantonese version of Community Integration Measures (CIM-C). The CIM is a client-centred questionnaire with 10 items; each item solicits a rating on a 5-point scale for a total score from 10 to 50. The CIM-C has demonstrated good internal consistency (Cronbach α, 0.84) and reliability (ICC, 0.84). A higher score indicates a higher level of community integration.
Community Integration Questionnaire (CIM) - followup | 12 weeks
  The level of community integration will be assessed by the Cantonese version of Community Integration Measures (CIM-C). The CIM is a client-centred questionnaire with 10 items; each item solicits a rating on a 5-point scale for a total score from 10 to 50. The CIM-C has demonstrated good internal consistency (Cronbach α, 0.84) and reliability (ICC, 0.84). A higher score indicates a higher level of community integration.
SATIS-Stroke - baseline | Baseline (0 week)
  The SATIS-Stroke will be used to evaluate the satisfaction with social participation among people with chronic stroke.The SATIS-Stroke contains 36 items using a four-point scale (0 to 3), with a maximum raw score of 108 (-5.11 to 5.08 in logits). The SATIS-Stroke has excellent internal consistency (Cronbach's α = 0.959) and good test-retest reliability (ICC = 0.91). A higher score indicates a high satisfaction level with social participation among people with chronic stroke.
SATIS-Stroke - midterm | 4 weeks
  The SATIS-Stroke will be used to evaluate the satisfaction with social participation among people with chronic stroke.The SATIS-Stroke contains 36 items using a four-point scale (0 to 3), with a maximum raw score of 108 (-5.11 to 5.08 in logits). The SATIS-Stroke has excellent internal consistency (Cronbach's α = 0.959) and good test-retest reliability (ICC = 0.91). A higher score indicates a high satisfaction level with social participation among people with chronic stroke.
SATIS-Stroke- post-training | 8 weeks
  The SATIS-Stroke will be used to evaluate the satisfaction with social participation among people with chronic stroke.The SATIS-Stroke contains 36 items using a four-point scale (0 to 3), with a maximum raw score of 108 (-5.11 to 5.08 in logits). The SATIS-Stroke has excellent internal consistency (Cronbach's α = 0.959) and good test-retest reliability (ICC = 0.91). A higher score indicates a high satisfaction level with social participation among people with chronic stroke.
SATIS-Stroke - followup | 12 weeks
  The SATIS-Stroke will be used to evaluate the satisfaction with social participation among people with chronic stroke.The SATIS-Stroke contains 36 items using a four-point scale (0 to 3), with a maximum raw score of 108 (-5.11 to 5.08 in logits). The SATIS-Stroke has excellent internal consistency (Cronbach's α = 0.959) and good test-retest reliability (ICC = 0.91). A higher score indicates a high satisfaction level with social participation among people with chronic stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Shamay Ng, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - The Hong Kong Polytechnic University, Hong Kong, Hong Kong
  - Shatin Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No